CLINICAL TRIAL: NCT01459120
Title: Comparing Door-to-door Versus Community Gathering in Providing HIV Counseling and Testing Within an Integrated Primary Health Care Package: a Cluster Randomized Trial in Rural Lesotho
Brief Title: Comparison of Door-to-door Versus Community Gathering to Provide HIV Counseling and Testing Services in Rural Lesotho
Acronym: DoDoPi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SolidarMed (Other)
Collaborators: Paray Mission Hospital, Thaba-Tseka (Unknown); Seboche Hospital, Botha-Bothe (Unknown)
Responsible Party: Principal Investigator, Niklaus Labhardt, Project Manager, SolidarMed
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DoDoPi-1
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: HIV/AIDS; Tuberculosis; Diabetes Mellitus; Arterial Hypertension
Keywords: Home-based HIV-testing; Voluntary Counseling and Testing; Community based testing; HIV/AIDS; Lesotho
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Diabetes Mellitus; Hypertension | interventions — Time-to-Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Door-to-Door (Experimental): Health care workers propose the integrated service package including VCT at the peoples' homes.
  Interventions: Other: Door-to-door
- Pitso (Active Comparator): Health care workers propose the integrated service package including VCT through community gatherings ("pitso").
  Interventions: Other: Pitso
- control (No Intervention): Within each cluster (catchment area of a health center), five villages are randomly chosen as comparators on cluster level. These villages get no particular intervention (VCT-campaign). However, routine services continue to be provided. These villages serve as a control for the third primary outcome that assesses the overall numbers newly enrolled into chronic HIV/AIDS care at facility-level.

INTERVENTIONS:
Other: Door-to-door — Health workers propose the integrated service package including VCT at the peoples' homes (home-based testing).
  Arms: Door-to-Door
Other: Pitso — Health care workers propose the integrated service package including VCT through community gatherings ("Pitso").
  Arms: Pitso

SUMMARY:
The purpose of this trial is to determine if door-to-door is more effective than community gathering in providing voluntary HIV counseling and testing (VCT) in communities in rural Lesotho. The voluntary HIV counseling and testing will be proposed as an integrated part of a package of proposed services. The package consists of: Blood-pressure measurement, blood-glucose measurement, Body-mass-index (adults), weight for height (children), catch-up vaccinations, deworming (children) Vitamin A (children & young women), family planning for eligible women, Tuberculosis screening and HIV counseling and testing.

DETAILED DESCRIPTION:
12 health centers (clusters) in rural Lesotho are matched according to their routine performance in VCT and enrollment into chronic HIV/AIDS care (average numbers tested positive and enrolled into HIV/AIDS care per month per facility). After matching, 6 health centers are randomly assigned to perform door-to-door VCT, whereas the others perform the traditional community gathering approach (called "pitso" in Sesotho). Within the catchment area of each health center five campaigns in five different, randomly selected villages, are held (one day VCT campaign per village). Within each cluster another five villages are randomly selected who do not get a particular campaign and serve as a control for each cluster. In each matched cluster-pair, both health centers conduct the five campaigns during the same week (one conducting it as door-to-door, the other one conducting it through "pitsos" (community gathering)).

Both approaches receive the same resources in terms of finances, time spending doing the VCT-campaign and human resources.

ELIGIBILITY:
Inclusion criteria:

* Not already known to be HIV-positive
* Resident in the catchment area of the health center where the campaign is conducted
* Provision of written informed consent to participate (signed by writing or fingerprint)
* In case of children: Provision of written informed consent by an adult care-taker

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proportion of newly tested HIV-positive clients over all clients tested for HIV during the campaigns
  Proportion refers to the proportion of newly tested HIV-positive clients among all clients tested for HIV during the voluntary counselling and testing campaigns in each arm.
Proportion of clients newly tested HIV-positive who enrolled into HIV/AIDS care within one month over all clients newly tested HIV-positive during the campaigns | 4 weeks after tested positive
  One month after the campaigns, enrollment of clients who newly tested HIV-positive at the campaign is assessed at the facilities based on the clinics' registers.
Overall number newly tested HIV-positive and enrolled into chronic HIV/AIDS-care at each facility | 4 weeks after campaign
  Between the two study-arms, the overall numbers will be compared in two ways:
  1. Total number positively tested and enrolled into care at the facility during the month after the campaign (this refers to the overall number at facility-level. Irrespective if these patients were tested during one of the campaigns or during routine activities at the facility)
  2. Total number positively tested and enrolled into care from the 5 villages where campaigns were held as compared to the five villages where no campaigns were held.
Absolute number of newly tested HIV-positive clients
  Refers to the overall number newly tested HIV-positive during the campaigns in both arms
Absolute number of clients newly tested HIV-positive who enrolled into HIV/AIDS care | 4 weeks after tested HIV-positive
  This refers to the absolute number newly tested HIV-positive during the campaigns who enrolled thereafter into chronic HIV/AIDS care within one month

SECONDARY OUTCOMES:
CD4-count among clients newly tested HIV-positive
  CD4-counts will be measured on site using a Point-of-care machine.
Clinical WHO-stage among clients newly tested HIV-positive
Proportion of clients screened positive for Tuberculosis during the campaigns
  All clients accessing services (irrespective of HIV-status) will be screened for TB by a nurse. Clients with a positive screening are provided sputum bottles and are entered in the Tuberculosis-suspect register.
Proportion of first-time HIV-testers among all clients accessing the testing services
Proportion of clients with positive tuberculosis screening who return 3 sputum-bottles within ≤ 5 days to the facility | 5 days after the campaign was held
  Tuberculosis-suspect registers and tuberculosis registers at the facility are used for verification
Proportion of clients with a positive Tuberculosis-screening who return their sputum-bottles and who have at least one AFB-positive smear. | 5 days after the campaign was held
  Tuberculosis suspect registers and Tuberculosis registers at the facility are used for verification.
Demographic characteristics of clients accessing the voluntary counseling and testing services
Absolute number of clients accessing the services at the campaigns who have a positive screening for Tuberculosis
Absolute number of clients with positive tuberculosis screening who return 3 sputum-bottles within ≤ 5 days to the facility | ≤ 5 days after the campaigns
Absolute number of clients with a positive Tuberculosis-screening who return their sputum-bottles and who have at least one AFB-positive smear. | ≤ 5 days after the campaign

CONTACTS AND LOCATIONS:
Overall Officials: Motlomelo Masetsibi, Principal Investigator — SolidarMed; Niklaus Labhardt, MD, MIH, Study Director — SolidarMed; Karolin Pfeiffer, MD, McommH, Study Chair — SolidarMed
Locations (2):
- Lesotho (2):
  - Seboche Hospital, Seboche, Botha-Bothe
  - Paray Hospital, Thaba-Tseka, Thaba-Tseka

REFERENCES:
- [Derived] Labhardt ND, Motlomelo M, Cerutti B, Pfeiffer K, Kamele M, Hobbins MA, Ehmer J. Home-based versus mobile clinic HIV testing and counseling in rural Lesotho: a cluster-randomized trial. PLoS Med. 2014 Dec 16;11(12):e1001768. doi: 10.1371/journal.pmed.1001768. eCollection 2014 Dec. PMID 25513807